CLINICAL TRIAL: NCT04977453
Title: A Phase 1/2, Open-label, Dose-escalation, and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Therapeutic Activity of GI-101 as a Single Agent and in Combination With Pembrolizumab, Lenvatinib or Local Radiotherapy in Patients With Advanced or Metastatic Solid Tumors (Keynote B59)
Brief Title: GI-101 as a Single Agent or in Combination With Pembrolizumab, Lenvatinib or Local Radiotherapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GI Innovation, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GII-101-P101 (MK-3475-B59); KEYNOTE-B59 (Other: Merck Sharpe and Dohme LLC)
Record Dates: First submitted 2021-07-09; First posted 2021-07-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Renal Cell Carcinoma; Urinary Bladder Cancer; Melanoma; Sarcoma; Microsatellite Stable Colorectal Carcinoma; Merkel Cell Carcinoma; Esophageal Squamous Cell Carcinoma; Cervical Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: GI-101/GI-101A; CD80-IgG4 Fc-IL2 variant; Immunotherapy; IL-2; Interleukin-2; Pembrolizumab; Lenvatinib; Radiotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Melanoma; Sarcoma; Carcinoma, Merkel Cell; Esophageal Squamous Cell Carcinoma; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- GI-101 (Experimental): Dose escalation: GI-101, multiple ascending doses
  Dose expansion:
  Interventions: Drug: GI-101
- GI-101 + Pembrolizumab (Experimental): Dose escalation: GI-101, multiple ascending doses
  Dose expansion:
  Interventions: Drug: GI-101; Drug: Pembrolizumab (KEYTRUDA®)
- GI-101 + Lenvatinib (Experimental): Dose optimization:
  Dose expansion:
  Interventions: Drug: GI-101; Drug: Lenvatinib
- GI-101 + Local Radiotherapy (Experimental): Dose optimization:
  Dose expansion:
  Interventions: Drug: GI-101; Radiation: Local Radiotherapy
- GI-101A (Experimental): Dose escalation: GI-101A, multiple ascending doses
  Dose expansion:
  Interventions: Drug: GI-101A
- GI-101A + Pembrolizumab (Experimental): Dose escalation: GI-101A, multiple ascending doses
  Dose expansion:
  Interventions: Drug: Pembrolizumab (KEYTRUDA®); Drug: GI-101A

INTERVENTIONS:
Drug: GI-101 — Recommended phase 2 dose of GI-101 will be administered via IV infusion Q3W up to 2 years (approximately 35 years).
  Arms: GI-101; GI-101 + Lenvatinib; GI-101 + Local Radiotherapy; GI-101 + Pembrolizumab
Drug: Pembrolizumab (KEYTRUDA®) — Pembrolizumab will be administered at a dose of 200 mg as IV infusion Q3W.
  Other Names: KEYTRUDA®
  Arms: GI-101 + Pembrolizumab; GI-101A + Pembrolizumab
Drug: Lenvatinib — Lenvatinib will be administered at an approved dose orally.
  Other Names: Lenvima®
  Arms: GI-101 + Lenvatinib
Radiation: Local Radiotherapy — Patients will receive SBRT prior to the first dose of GI-101
  Arms: GI-101 + Local Radiotherapy
Drug: GI-101A — Recommended phase 2 dose of GI-101A will be administered via IV infusion Q3W up to 2 years (approximately 35 years).
  Arms: GI-101A; GI-101A + Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and therapeutic activity of GI-101/GI-101A as a single agent or in combination with pembrolizumab, lenvatinib or local radiotherapy (RT) over a range of advanced and/or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, dose-escalation and expansion study to evaluate the safety, tolerability and anti-tumor effect of GI-101/GI-101A as a single agent or in combination with pembrolizumab, lenvatinib or local RT over a range of advanced and/or metastatic solid tumors.

This study will comprise six parts.

* Part A: Dose-escalation and expansion cohorts of GI-101 monotherapy
* Part B: Dose-escalation and expansion cohorts of GI-101 plus pembrolizumab
* Part C: Dose-optimization and expansion cohorts of GI-101 plus lenvatinib
* Part D: Dose-optimization and expansion cohorts of GI-101 plus local RT
* Part E: Dose-escalation and expansion cohorts of GI-101A monotherapy
* Part F: Dose-escalation and expansion cohorts of GI-101A plus pembrolizumab

GI-101/GI-101A is a novel bi-specific Fc fusion protein containing the CD80 ectodomain as an N-terminal moiety and an interleukin (IL)-2 variant as a C-terminal moiety configurated via a human immunoglobulin G4 (IgG4) Fc.

GI-101A is an abbreviation of advanced GI-101 with an improved formulation for manufacture consistency.

Drug Information available for: Pembrolizumab (https://www.keytrudahcp.com), Lenvatinib (http://www.lenvima.com)

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females aged ≥ 18 years (or ≥ 19 years according to local regulatory guidelines) at the time of screening.
* Has adequate organ and marrow function as defined in protocol.
* Measurable disease as per RECIST v1.1.
* ECOG performance status 0-1.
* Adverse events related to any prior chemotherapy, radiotherapy, immunotherapy, other prior systemic anti-cancer therapy, or surgery must have resolved to Grade ≤1, except alopecia and Grade 2 peripheral neuropathy.
* HIV infected patients must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease as defined in protocol.

Key Exclusion Criteria:

* Has known active CNS metastases and/or carcinomatous meningitis.
* An active second malignancy
* Has active or a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has active tuberculosis or has a known history of active tuberculosis
* Active or uncontrolled infections, or severe infection within 4 weeks before study treatment administration.
* History of chronic liver disease or evidence of hepatic cirrhosis, except patients with liver metastasis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Previous immunotherapies related to mode of action of GI-101.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive medications within 2 weeks prior to Cycle 1 Day 1.
* Administration of prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment.
* Radiotherapy within the last 2 weeks before start of study treatment administration, with exception of limited field palliative radiotherapy (except Part D).
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1.
* Known hypersensitivity to any of the components of the drug products and/or excipients of GI-101, pembrolizumab or lenvatinib.

Other protocol defined inclusion exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of Dose-Limiting Toxicity (DLTs) | Study Day 1, assessed up to approximately 24 months
  Based on toxicities observed.
Incidence, nature, and severity of adverse events (AEs) and immune-related AEs (irAEs) | Study Day 1, assessed up to approximately 24 months
  Based on toxicities observed.
Objective Response Rate (ORR) according to RECIST version 1.1 | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of GI-101/GI-101A | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Half-life of GI-101/GI-101A (T1/2) | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Area under the plasma concentration versus time curve (AUC) of GI-101/GI-101A | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Disease control rate (DCR) according to RECIST version 1.1 | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.
Duration of objective Response (DoR) according to RECIST version 1.1 | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.
Time to Tumor Response (TTR) according to RECIST version 1.1 | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.
Progression-Free Survival (PFS) according to RECIST version 1.1 | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.
ORR per iRECIST guidelines | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.
DCR per iRECIST guidelines | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging.

OTHER OUTCOMES:
Incidence of anti-GI-101/GI-101A antibody (ADA) and neutralizing antibody (Nab) | Study Day 1, assessed up to approximately 24 months
  Serum will be assessed for the presence of ADA and Nab based on the appropriate assay.
Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry at various time points | Study Day 1, assessed up to approximately 24 months
  Peripheral immune cell subpopulation (e.g., CD4+ T cells, CD8+ T cells, regulatory T cells) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Nari Yun, PhD, Study Director — GI Innovation
Locations (7):
- United States (2):
  - Tisch Cancer Institute (TCI), Icahn School of Medicine, New York, New York
  - Carolina Biooncology Institute, Huntersville, North Carolina
- South Korea (5):
  - Chungnam National University Hospital, Daejeon, Daejeon
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Kyeonggi-do
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No